CLINICAL TRIAL: NCT03109808
Title: Impact of a Personalized Video in Oral Hygiene Motivation
Acronym: GOPERIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: University of Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16/065
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-02

CONDITIONS: Dental Hygiene

STUDY DESIGN:
Intervention Model Description: * Allocation : Randomized (with stratification on center and gender)
  * Endpoint Classification : Safety/Efficacy Study
  * Intervention Model : Parallel Assignment
  * Masking : Double blind (Operator, Outcomes Assessor)
  * Primary Purpose : Prevention
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-health strategy (Experimental): Assigned intervention: e-health strategy
  Interventions: Other: e-health strategy
- Traditional Oral Hygiene Education (Active Comparator): Assigned intervention: traditional oral hygiene education
  Interventions: Other: Traditional Oral Hygiene Education

INTERVENTIONS:
Other: e-health strategy — * First, a personalized video of the patient's oral hygiene routine (toothbrushing and interdental hygiene) is recorded and made available to him-her via a cloud-based system. The patient is instructed to view it with his-her smartphone and/or tablet when brushing his-her teeth.
  * Second, the patient is registered in a text-based recall system. This recall system will remind him-her the oral hygiene regimen suited to his-her personal situation and contains a link to his cloud-hosted video. 12 text messages for each patient will be sent over the course of the study (8 weeks). This is a two-way system as patients will be inquired about their compliance to oral hygiene. If the patient declare compliance, he-she will be congratulated (positive reinforcement). If the patient declares non-compliance, he-she will be informed he-she will be offered additional counselling at the next appointment.
  Arms: e-health strategy
Other: Traditional Oral Hygiene Education — traditional oral hygiene education
  Arms: Traditional Oral Hygiene Education

SUMMARY:
Impact of a personalized video in oral hygiene motivation: The study hypothesis is that the use of a personalized oral hygiene video, made available to the patient via a cloud-based system, in conjunction with a text-based two-way recall system will increase patient compliance, hence leading to improvement or oral hygiene.

DETAILED DESCRIPTION:
The strategy studied is composite:

* First, a personalized video of the patient's oral hygiene routine (toothbrushing and interdental hygiene) is recorded and made available to him-her via a cloud-based system. The patient is instructed to view it with his-her smartphone and/or tablet when brushing his-her teeth.
* Second, the patient is registered in a text-based recall system. This recall system will remind him-her the oral hygiene regimen suited to his-her personal situation and contains a link to his cloud-hosted video. 12 text messages for each patient will be sent over the course of the study (8 weeks). This is a two-way system as patients will be inquired about their compliance to oral hygiene. If the patient declare compliance, he-she will be congratulated (positive reinforcement). If the patient declares non-compliance, he-she will be informed he-she will be offered additional counselling at the next appointment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older, having a good understanding of French language (read, write, speak, listen)
* With at least 20 teeth, including 4 first molars and 4 first or second premolars (4 interdental sites between premolars and molars)
* Patient attending an appointment in a centre participating to the trial
* Patient able to support treatment
* Patient affiliated to a health insurance scheme
* Patient giving his informed consent and accepting the modalities of the study
* Patient agreeing to attend up to 4 appointments dedicated to the study, during 8 weeks after the initial appointment (motivational interview)
* Patient in possession of an internet-enabled smartphone or tablet
* Patient has a personal e-mail address
* Patient agreeing to be registered within the system of text-based recalls for the duration of the study

Exclusion Criteria:

* Patient having previously benefited from a periodontal therapy (less than 1 year ago) or currently enrolled in a periodontal therapy program
* Patient having previously benefited from an oral hygiene motivation session less than 1 year ago
* Patient has had a calculus removal procedure less than 1 month ago
* Patient bears orthodontic appliances (any kind, for 1 or both arches)
* Patient bears removable dental prosthesis (any kind, for 1 or both arches)
* Patient allergic to benzoic acid preservatives (or thought to be)
* Patient has a high risk of infective endocarditis
* Patient benefiting from antiaggregant or anticoagulation therapy
* Patient is haemophilic
* Patient is unable to answer questions
* Patient is unable (from a cognitive or physical standpoint) to perform toothbrushing twice a day
* Patient is unable (from a cognitive or physical standpoint) to use interdental brushes and/or dental floss (at least once a day)
* Patient uses on a regular basis (more than once a week) interdental brushes and/or dental floss in addition to toothbrushing
* Patient under tutelage or guardianship
* Patient deaf or blind
* Non cooperative patient
* Patient will be changing geographical location (ie. moving away) during the duration of the study, hence compromising follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-02-15 (Estimated); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
O'Leary Plaque Control Record | 8 weeks
  Measures the presence (1) or absence (0) of dental plaque on 6 sites per tooth for all teeth in mouth

SECONDARY OUTCOMES:
Bleeding on Probing Index | 8 weeks
  Measures the presence (1) or absence (0) of bleeding at the gingival margin up to 30 seconds after the insertion of the periodontal probe in the sulcus
Patient satisfaction | 8 weeks
  Measured by a dedicated questionnaire
Patient motivation | 8 weeks
  Measured by a dedicated questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Liege, Liège, Belgium
- Hospices Civils de Lyon - Service de Consultations et de Traitements Dentaires, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garyga V, Pochelu F, Thivichon-Prince B, Aouini W, Santamaria J, Lambert F, Maucort-Boulch D, Gueyffier F, Gritsch K, Grosgogeat B. GoPerio - impact of a personalized video and an automated two-way text-messaging system in oral hygiene motivation: study protocol for a randomized controlled trial. Trials. 2019 Dec 10;20(1):699. doi: 10.1186/s13063-019-3738-0. PMID 31823812